CLINICAL TRIAL: NCT01902368
Title: A Prospective Trial of Celiac Disease Screening
Brief Title: Celiac Disease Screening
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding was obtained.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Leffler, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 2012P000326
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Celiac Disease
Keywords: Gluten free diet
MeSH Terms: conditions — Celiac Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- screen detected, early diagnosis cohort (Other): Subjects will be informed they have celiac disease and will be started on the gluten free diet.
  Interventions: Other: gluten free diet
- screen detected, delayed diagnosis cohort (No Intervention): Subjects will not be told they have celiac disease and will not start the gluten free diet.

INTERVENTIONS:
Other: gluten free diet
  Arms: screen detected, early diagnosis cohort

SUMMARY:
The purpose of this study is to see if it makes sense to test people for celiac disease who have a first or second degree relative (parent, sibling, child, grandparent, aunt or uncle) with celiac disease. The investigators will check to see what differences there are in the health and quality of life between those who know they have celiac disease and start the gluten free diet and those who do not.

DETAILED DESCRIPTION:
Our overall hypothesis is that first and second degree relatives of individuals with celiac disease benefit from screening and diagnosis of celiac disease. Secondary hypotheses are:

1. The number needed to test and cost to benefit one person though celiac disease screening are within acceptable ranges of 33 tested and < $10,000 spent.
2. Treatment does not lead to adverse metabolic changes.
3. Intestinal biopsy is unnecessary for accurate diagnosis in a substantial subset of adults.

Aim 1. Determine the effect of screen detected celiac disease on health related quality of life.

* Evaluate change in health related quality of life at one year in participants randomized to the screen detected, early diagnosis cohort compared to the screen detected, delayed diagnosis, clinically detected and non-celiac control cohorts.
* Evaluate change in symptoms, psychological well-being and burden of treatment at one year in the screen detected, early diagnosis cohort compared to the screen detected, delayed diagnosis, clinically detected and non-celiac control cohorts.
* Evaluate the cost per diagnosis and the number needed to test for the diagnosis of individuals who will have a clinically meaningful improvement in health related quality of life attributable to treatment of celiac disease.

Aim 2: Assess the effect of screen detected celiac disease on nutritional and metabolic indices.

* Compare changes bone density, body mass index, Reynolds Cardiovascular Risk Score, and nutritional indices at one year in the screen detected, early diagnosis cohort compared to the screen detected, delayed diagnosis, clinically detected and non-celiac control cohorts.

Aim 3: Evaluate the reliability of using serologic tests in combination with intestinal fatty acid binding protein vs. intestinal biopsy to confirm celiac disease diagnosis in adults.

* Prospectively assess the sensitivity and specificity of a novel non-invasive celiac diagnostic algorithm in comparison to the current gold standard of small intestinal biopsy histology.
* Model the cost of modified, non-invasive celiac testing vs. classical testing with endoscopic biopsy in both screen-detected and clinically identified celiac disease.

ELIGIBILITY:
Inclusion Criteria:

* Be ambulatory, community dwelling, 18 to 80 years, inclusive
* For the screening cohort:

  * Have a first or second degree family member with known biopsy-proven celiac disease.
  * Have not been on a gluten-free diet in the past 6 months
  * Have not received a prior diagnosis of celiac disease at any time
* For the clinically detected cohort

  * Have biopsy proven celiac disease detected based on clinical symptoms and on a gluten free diet for less than 1 month.

Exclusion Criteria:

* For the screen detected cohort, have significantly severe symptoms (as judged by the investigator) at screening which preclude randomization;
* Be on a gluten-free diet or have been on a gluten-free diet within the past 6 months.
* Be pregnant or planning pregnancy in the study time period
* Be taking corticosteroids or immunomodulators
* Have a history of significant concomitant gastrointestinal disease or other comorbidity judged by the investigator to potentially interfere with study outcomes
* Be unable or unwilling to cooperate with the study protocol
* Have insufficient knowledge of English to complete study surveys

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
change in health related quality of life | Baseline, 3, 6, 9 and 12 months
  as measured by the EQ-5D

SECONDARY OUTCOMES:
change in celiac symptoms | Baseline, 3, 6, 9 and 12 months
  as measured by the Celiac Symptom Index
change in bone density | Baseline and 12 months
  as measured by dual energy x-ray absorptiometry
change in psychological well-being | Baseline, 3, 6, 9, and 12 months
  as measured by the Psychological General Well-Being Index
change in burden of treatment | baseline, 3, 6, 9, and 12 months
  as measured by the disease burden visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Leffler, MD, MS, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States